CLINICAL TRIAL: NCT03778983
Title: Cognitive Development After Pediatric Liver Transplantation
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CDPLT
Record Dates: First submitted 2018-11-13; First posted 2018-12-19 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Cognitive Development After Pediatric Live Transplantation
Keywords: Cognitive Development; Pediatric Live Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Live Transplantation Group: Children who underwent pediatric Ltx at RenJi Hospital before 12 month, and now age between 2 and 7 years;

SUMMARY:
The purpose of this study is to investigate the cognitive performance after pediatric live transplantation.

DETAILED DESCRIPTION:
During the last 20 years, survival rates after pediatric liver transplantation (Ltx) have increased steadily. Today, pediatric Ltx is a well-established treatment for a variety of liver diseases in their final stage. Even in relative indications (i.e. certain metabolic diseases), liver transplantation is a promising treatment option that actually is becoming increasingly important in clinical practice .

Importantly, childhood cognitive ability is highly predictive for educational achievement and later occupational outcomes as well as health behavior . Current research indicates that liver transplanted children are at higher risk for developing cognitive deficits compared to the age-matched normal population .

The aim of present study is to evaluate the cognitive development after pediatric liver transplantation. The investigators expect to understand of the association between cognitive deficits and certain disease-related variables, which may be contribute to optimizing clinical care of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients accepted Live Transplantation before 12 month, and now age between 2 and 7 years;
2. residency in China;
3. sufficient Chinese language skills;
4. at least 1 year post-Ltx;
5. no acute diseases;
6. no mental handicap.

Exclusion Criteria:

1. Re-transplantation
2. Patients with localized or systemic infection
3. Patients cor-morbid with auto-immune disease
4. Combined liver and kidney transplantation
5. Lack of informed consent

Ages: 2 Years to 7 Years | Sex: All
Age Groups: Child
Gender Based: Yes — Chinese
Study Population: The study chooses children who underwent pediatric Ltx before 12 month at RenJi Hospital , Chinese, now age before 2 and 7 years . Inclusion criteria were as follows: (1) age between2 and7 years, (2) residency in China, (3) sufficient Chinese language skills, (4) at least 1 year post-Ltx, (5) no acute diseases and (6) no mental handicap.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Intelligence function evaluated by Wechsler Intelligence Scale IV | at least 1 year after pediatric live transplantation
  Wechsler Intelligence Scale IV (WISC-IV) is the newly released and completely revised Chineseversion of the Wechsler Intelligence Scale for Children-fourth edition(WISC-IV) . A global intelligence score, the Total IQ, is comprised of four index scores: (i) Verbal Comprehension Index, which includes the subtests Similarities, Vocabulary and Comprehension; (ii) Perceptual Reasoning Index, which consists of Block Design, Picture Concepts and Matrix Reasoning; (iii) Working Memory Index, which encompasses the subtests Digit Span and Letter Number Sequencing; (iv) Processing Speed Index, which is composed of the subtests Coding and Symbol Search. The normative populations mean (M) is 100, and the standard deviation (SD) is 15 for all indices.The lower the intelligence score, the worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, MD, Study Chair — Anesthesiology Department Renji Hospital, Shanghai
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China